CLINICAL TRIAL: NCT01561534
Title: Long-term Results of Mandibular/Maxillary Reconstruction With Vascularized Free Fibula Flap and Computer-guided Implant Surgery
Brief Title: Vascularized Free Fibula Flap and Computer-guided Implant Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, MICHELE DE BENEDITTIS, principal investigator, University of Bari
Other Study IDs: 0104
Record Dates: First submitted 2012-03-13; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Oral Tumor
Keywords: fibula flap; oral implants; computer-guided
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The rehabilitation of patients affected by defects of the jaws after tumor resection is still very challenging. Resection can lead to significant facial deformity, impaired oral functions such as speech, swallowing, saliva retention, and concomitant psychological problems. Moreover, the loss of teeth and the alveolar and basal jawbone can lead to significant impairment of mastication. The reconstruction of such defects with autogenous bone grafts or revascularized free flaps has become a valuable means for the rehabilitation of these patients. Major benefits of such procedure include an usually low morbidity of the donor site and an extensive length of the bone graft. Moreover, vascularized grafts provide a good bulk of bone in which to place implants and a satisfactory contour. In fact, after reconstruction, local hard and soft tissue conditions often exclude the integration of conventional dentures because of the impairment of dental prosthetic retention by thin cutaneous tissue, the thickness of subcutaneous tissues, the absence of a perilingual and vestibular groove, and the fragility of soft tissues. In Literature it has been well established the high biologic value of vascularized fibula grafts regarding the potential of implant osseointegration, which seemed to be equal to regional mandibular or maxillary bone and eventually capable to provide sufficient stabilization of prosthesis.

It must be kept in mind that the final prosthetic success may be affected by some difficulties in this clinical scenario. These include the limited opening of the scar-contracted oral cavity, the huge amount of soft tissue covering the fibula, with little information about the profile of the underlying harvested bone, the need for limited bony exposure in a field that may well have been irradiated and they all may cause poor prosthetically-guided implant positioning and eventually disappointing results in dental rehabilitation, either functionally or esthetically. It can be postulated that these complications can be overcome, or at least reduced, by adopting the new methods of computed tomography (CT)-assisted implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with free fibula flaps for maxillary and mandibular reconstruction needing full arch or quasi full arch rehabilitation

Exclusion Criteria:

* radiation therapy
* malignant tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with free fibula flaps for maxillary and mandibular reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
change of peri-implant bone level from baseline at 12 and 24 months | 12 months and 24 months
  successful implants will be those with peri-implant bone resorption less than 1.5 mm in the first year of function and less than
  0.2 mm in the subsequent years

SECONDARY OUTCOMES:
pain | 12 months and 24 months
peri-implant infection | 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MICHELE DE BENEDITTIS, RESEARCHER, Principal Investigator — University of Bari
Locations (1):
- Ospedale regionale F. Miulli, Acquaviva delle Fonti, Bari, Italy